CLINICAL TRIAL: NCT02029625
Title: A Clinical Trial to Compare the Pharmacokinetics and Safety of NVP-1205 and Coadministration of Rosuvastatin and Ezetimibe in Healthy Male Volunteers
Brief Title: Compare the Pharmacokinetics of NVP-1205 and Coadministration of Rosuvastatin and Ezetimibe
Acronym: NVP-1205
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: NVP-1205-01
Record Dates: First submitted 2014-01-05; First posted 2014-01-08 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVP-1205 (Experimental): administration of NVP-1205(rosuvastatin+ezetimibe)
  Interventions: Drug: NVP-1205
- rosuvastatin and ezetimibe (Active Comparator): coadministration of rosuvastatin and ezetimibe
  Interventions: Drug: rosuvastatin and ezetimibe

INTERVENTIONS:
Drug: NVP-1205 — rosuvastatin/ezetimibe fixed dose combination orally, once daily on Period 1 or Period 2
  Other Names: NVP-1205(rosuvastatin+ezetimibe)
  Arms: NVP-1205
Drug: rosuvastatin and ezetimibe — coadministration of rosuvastatin and ezetimibe orally, once daily on Period 1 or Period 2
  Other Names: Crestor and Ezetrol
  Arms: rosuvastatin and ezetimibe

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of NVP-1205 and coadministration of rosuvastatin and ezetimibe.

DETAILED DESCRIPTION:
rosuvastatin and ezetimibe(anti-dyslipidemia)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age between 19 and 55 signed informed consent

Exclusion Criteria:

* subjects have a history of allergy reaction of this drug or other drugs

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
AUClast | 0-96hr

SECONDARY OUTCOMES:
AUCinf | 0-96hr

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Yo Ran, M.D., Ph,D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National Hospital, Jung-gu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No